CLINICAL TRIAL: NCT03285178
Title: A Randomized, Placebo-controlled, Phase 2 Study to Evaluate the Safety and Pharmacodynamics of Once-daily Oral IW-1701 in Patients With Stable Sickle Cell Disease
Brief Title: A Study of the Effect of IW-1701 (Olinciguat), a Stimulator of Soluble Guanylate Cyclase (sGC), on Patients With Sickle Cell Disease (SCD)
Acronym: STRONG SCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1701-202
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; SCD; Olinciguat; IW-1701
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- IW-1701 (Olinciguat) 2 mg (Experimental): After a single-blind treatment with placebo once daily (QD) for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1, participants received 1 mg olinciguat QD Week 1 and 2 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
  Interventions: Drug: IW-1701
- IW-1701 (Olinciguat) 4 mg (Experimental): After a single-blind treatment with placebo QD for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1, participants received 2 mg olinciguat QD Week 1 and 4 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
  Interventions: Drug: IW-1701
- IW-1701 (Olinciguat) 6 mg (Experimental): After a single-blind treatment with placebo QD for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1, participants received 3 mg olinciguat QD Week 1 and 6 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
  Interventions: Drug: IW-1701
- IW-1701 (Olinciguat) 18 mg (Experimental): After a single-blind treatment with placebo QD for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1, participants received 6 mg olinciguat QD Days 1-7, 12 mg olinciguat QD Weeks 1-3, and 18 mg olinciguat QD Weeks 4-12 under protocol Amendment 4 and later.
  Interventions: Drug: IW-1701
- Placebo (Placebo Comparator): After a single-blind treatment with placebo QD for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1, participants received placebo treatment QD for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-1701 — Oral Tablet
  Other Names: Olinciguat
  Arms: IW-1701 (Olinciguat) 18 mg; IW-1701 (Olinciguat) 2 mg; IW-1701 (Olinciguat) 4 mg; IW-1701 (Olinciguat) 6 mg
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
The primary objective of the 1701-202 STRONG SCD study is to evaluate the safety and tolerability of different dose levels of IW-1701 compared with placebo when administered daily for approximately 12 weeks to patients with stable SCD. Exploratory objectives include evaluation of pharmacokinetic (PK) as well as evaluation of the effect of IW-1701 on symptoms of SCD, health-related quality of life, and biomarkers of pharmacodynamic (PD) activity.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patient is ambulatory male or female 16 to 70 years of age at the Screening Visit.
2. Patient has SCD, including homozygous hemoglobin S (HbSS), hemoglobin SC disease (HbSC), heterozygous hemoglobin S-beta zero (HbSβ0)-thalassemia, or heterozygous hemoglobin S-beta plus (HbSβ+)-thalassemia, documented in their medical history.
3. If patient is on medication(s) for SCD, such as hydroxyurea (HU), are on a stable regimen.
4. Per medical history and/or patient recall, patient has had at least 1 and no more than 10 sickle cell-related pain crises in the 12 months before the Screening Visit and none occurring in the 4 weeks before the Randomization Visit.
5. Patient completes daily eDiary entries for at least 10 days during the last 14 days of the Run in Period as assessed at the Randomization Visit.
6. Women of childbearing potential must have a negative pregnancy test prior to randomization and must agree to use protocol-specified contraception from the Screening Visit through 90 days after the final dose of study drug.
7. Male patients must be surgically sterile by vasectomy (conducted ≥60 days before the Screening Visit or confirmed via sperm analysis) or must agree to use protocol-specified contraception and agree to refrain from sperm donation from the Screening Visit through 90 days after the final dose of study drug.

EXCLUSION CRITERIA

1. Patient requires a program of prescheduled, regularly administered chronic blood transfusion therapy.
2. Patient has been hospitalized for an SCD-related complication in the 4 weeks before the Randomization Visit.
3. Patient has taken opioid(s) >200 morphine mg equivalent/day within the 4 weeks before the Randomization Visit.
4. Patient is taking aspirin ≥325 mg daily, P2Y12 inhibitors, any anticoagulant medication, specific inhibitors of phosphodiesterase 5 (PDE5), nonspecific inhibitors of phosphodiesterase 5 (PDE5), moderate or strong cytochrome P450 3A (CYP3A) inhibitors, any supplements for the treatment of erectile dysfunction, riociguat, or nitrates or nitric oxide donors in any form.
5. Patient has major concurrent illness or medical condition that in the opinion of the Investigator would preclude participation in a clinical study.

NOTE: Other inclusion and exclusion criteria apply, per protocol

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (30):
  - Children's Hospital of Orange County, Orange, California
  - MedStar Health Research Institute, MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Howard University Center for Sickle Cell Disease, Washington D.C., District of Columbia
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - Century Clinical Research, Inc., Fort Lauderdale, Florida
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins School of Medicine Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan-Detroit, Detroit, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Hackensack University Medical Center, Pediatric Hematology and Oncology, Hackensack, New Jersey
  - Jacobi Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - East Carolina University - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - East Carolina University Brody School of Medicine, Department of Pediatrics, Division of Pediatric Hematology, Greenville, North Carolina
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - The Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Accurate Clinical Research, Baytown, Texas
  - "UT Health Clinical Research Unit Center for Clinical and Translational Sciences, Houston, Texas
  - Mays Cancer Center UT Health San Antonio, San Antonio, Texas
  - Virginia Commonwealth University - Clinical Research Unit, Richmond, Virginia
  - Blood Center of Wisconsin (BCW), Wauwatosa, Wisconsin
- Lebanon (2):
  - Hammoud Hospital University Medical Center, Sidon
  - Nini Hospital, Tripoli
- United Kingdom (5):
  - Royal London Hospital, London
  - Whittington Hospital, London
  - Guys and St Thomas NHS Foundation Trust - Evelina London Childrens Hospital, London
  - Guy's Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a 2-week single-blind placebo Run-in, eligible participants were stratified by hydroxyurea (hydroxycarbamide [HU]) use (yes or no) and randomly assigned to double-blind study drug (olinciguat or placebo).
  * Under Amendment 3 and earlier: Participants were assigned in a 1:1:1:1 ratio to placebo, 2 mg olinciguat, 4 mg olinciguat, or 6 mg olinciguat.
  * Under Amendment 4 and later: Participants were assigned in a 3:1 ratio to 18 mg olinciguat or placebo.
Groups:
- Single-Blind Run-in: Placebo: Single-blind treatment with placebo once daily (QD) for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1.
- Double-Blind Treatment: Placebo 1: Participants received placebo treatment QD for 12 weeks under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
- Double-Blind Treatment: Placebo 2: Participants received placebo treatment QD for 12 weeks under protocol Amendment 4 and later.
- Double-Blind Treatment: IW-1701 (Olinciguat) 2 mg: Participants received 1 mg olinciguat QD Week 1 and 2 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
- Double-Blind Treatment: IW-1701 (Olinciguat) 4 mg: Participants received 2 mg olinciguat QD Week 1 and 4 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
- Double-Blind Treatment: IW-1701 (Olinciguat) 6 mg: Participants received 3 mg olinciguat QD Week 1 and 6 mg olinciguat QD Weeks 2-12 under the original protocol, Amendment 1, Amendment 2, and Amendment 3.
- Double-Blind Treatment: IW-1701 (Olinciguat) 18 mg: Participants received 6 mg olinciguat QD Days 1-7, 12 mg olinciguat QD Weeks 1-3, and 18 mg olinciguat QD Weeks 4-12 under protocol Amendment 4 and later.
Period: Single-Blind Run-In Period
Arm/Group | Single-Blind Run-in: Placebo | Double-Blind Treatment: Placebo 1 | Double-Blind Treatment: Placebo 2 | Double-Blind Treatment: IW-1701 (Olinciguat) 2 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 4 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 6 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 18 mg
Started | 88 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 70 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Pandemic Precautions - Suspended by Institutional Review Board (IRB) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Pandemic Precautions- Suspended per Local Guidelines | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Single-Blind Run-in: Placebo | Double-Blind Treatment: Placebo 1 | Double-Blind Treatment: Placebo 2 | Double-Blind Treatment: IW-1701 (Olinciguat) 2 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 4 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 6 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 18 mg
Started | 0 | 10 | 9 | 8 | 8 | 11 | 24
Completed | 0 | 8 | 6 | 7 | 6 | 9 | 21
Not Completed | 0 | 2 | 3 | 1 | 2 | 2 | 3
Not completed — Randomized Mistakenly During the Run-In Period - Did Not Receive Study Drug | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 2 | 1
Not completed — COVID-19 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Treatment: Placebo 1 | Double-Blind Treatment: Placebo 2 | Double-Blind Treatment: IW-1701 (Olinciguat) 2 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 4 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 6 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 18 mg | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 11 | 24 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (9.43) | 31.5 (9.29) | 26.3 (10.51) | 34.5 (11.38) | 34.4 (13.34) | 32.7 (12.63) | 32.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 7 | 6 | 14 | 44
  Male | 2 | 3 | 3 | 1 | 5 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 4 | 8 | 8 | 10 | 15 | 53
  White | 0 | 4 | 0 | 0 | 0 | 9 | 13
  Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 7 | 6 | 8 | 10 | 22 | 60
  Not Reported | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Unknown | 1 | 0 | 1 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Treatment: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. A serious AE (SAE) is defined as any AE occurring at any dose that results in any of the following: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; other important medical event. A TEAE is an event that occurs after initiation of randomized study drug through 28 days after study drug discontinuation. Events were categorized by grade: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death, and as related or unrelated to study drug. Adverse Events of special interest (AESIs) included symptomatic or Grade ≥2 hypotensive events and/or tachycardia AEs, bleeding events, pulmonary edema, and bone-related events, including fractures.
Time Frame: First dose of randomized drug through 28 days after study drug discontinuation. Median number of weeks of treatment was 12.30, 11.85, 12.20, 12.20, 12.10, and 12.10, respectively, for Placebo 1, Placebo 2, Olinciguat 2 mg, 4 mg, 6 mg, and 18 mg groups.
Population: Safety Population: Randomized participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Treatment: Placebo 1 | Double-Blind Treatment: Placebo 2 | Double-Blind Treatment: IW-1701 (Olinciguat) 2 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 4 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 6 mg | Double-Blind Treatment: IW-1701 (Olinciguat) 18 mg
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 11 | 24
Participants
  Participants with >=1 TEAE | 6 | 6 | 5 | 5 | 8 | 21
  Participants with >=1 Grade 3-5 TEAE | 2 | 2 | 2 | 3 | 4 | 7
  Participants with >=1 Study Drug-Related TEAE | 3 | 0 | 2 | 0 | 4 | 7
  Participants with >=1 SAE | 2 | 1 | 2 | 3 | 4 | 6
  Participants with >=1 TEAE Leading to Study Drug Discontinuation | 0 | 0 | 0 | 0 | 0 | 2
  Participants with >=1 AESI | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Double-Blind Treatment: Number of TEAE Events
Description: An AE is any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any AE occurring at any dose that results in any of the following: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; other important medical event. A TEAE is an event that occurs after initiation of randomized study drug through 28 days after study drug discontinuation. Events were categorized by grade: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death, and as related or unrelated to study drug. If a participant had more than 1 occurrence in the same event category, only the occurrence with closest relationship to study drug was counted.
Time Frame: as for outcome 1
Population: Safety Population: Randomized participants who received at least 1 dose of study drug. Participants with >=1 TEAE.
Measure: Number; unit: TEAE Events
Groups:
- Placebo 1; IW-1701 (Olinciguat) 2 mg; IW-1701 (Olinciguat) 4 mg; IW-1701 (Olinciguat) 6 mg: Participants receiving treatment under the original protocol, Amendment 1, Amendment 2, and Amendment 3
- Placebo 2; IW-1701 (Olinciguat) 18 mg: Participants receiving treatment under protocol Amendment 4 and later
Arm/Group | Placebo 1 | Placebo 2 | IW-1701 (Olinciguat) 2 mg | IW-1701 (Olinciguat) 4 mg | IW-1701 (Olinciguat) 6 mg | IW-1701 (Olinciguat) 18 mg
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 8 | 21
TEAE Events | 26 | 29 | 36 | 30 | 39 | 101

3. Primary Outcome: Double-Blind Treatment: Number of Participants With ≥1 TEAE, by Maximum Severity
Description: An AE is any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any AE occurring at any dose that results in any of the following: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; other important medical event. A TEAE is an event that occurs after initiation of randomized study drug through 28 days after study drug discontinuation. Events were categorized by grade: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death, and as related or unrelated to study drug. If a participant had more than 1 occurrence in the same event category, only the most severe occurrence was counted.
Time Frame: as for outcome 1
Population: Safety Population: Randomized participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- IW-1701 (Olinciguat) 4 mg: Participants receiving treatment under the original protocol, Amendment 1, Amendment 2, and Amendment 3I
Arm/Group | Placebo 1 | Placebo 2 | IW-1701 (Olinciguat) 2 mg | IW-1701 (Olinciguat) 4 mg | IW-1701 (Olinciguat) 6 mg | IW-1701 (Olinciguat) 18 mg
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 11 | 24
Participants
  Participants with ≥1 TEAE: Any | 6 | 6 | 5 | 5 | 8 | 21
  Participants with ≥1 TEAE: Grade 1 | 0 | 4 | 0 | 2 | 2 | 6
  Participants with ≥1 TEAE: Grade 2 | 4 | 0 | 3 | 0 | 2 | 8
  Participants with ≥1 TEAE: Grade 3 | 2 | 2 | 2 | 3 | 4 | 7
  Participants with ≥1 TEAE: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with ≥1 TEAE: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Double-Blind Treatment: Number of Participants With Study Drug-Related TEAEs
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Safety Population: Randomized participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo 1 | Placebo 2 | IW-1701 (Olinciguat) 2 mg | IW-1701 (Olinciguat) 4 mg | IW-1701 (Olinciguat) 6 mg | IW-1701 (Olinciguat) 18 mg
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 11 | 24
Participants | 3 | 0 | 2 | 0 | 4 | 7

ADVERSE EVENTS:
Time Frame: AEs during Single-blind Run-in Period were collected from first dose of Run-in placebo up to the first dose of randomized study drug, up to 17 days. AEs during the Double-Blind Period: First dose of randomized drug through 28 days after study drug discontinuation. Median number of weeks of treatment was 12.30, 11.85, 12.20, 12.20, 12.10, and 12.10, respectively, for Placebo 1, Placebo 2, Olinciguat 2 mg, 4 mg, 6 mg, and 18 mg groups.
Description: All Cause mortality was collected for the duration of the study, mean 141.2 days.
Groups:
- Single-Blind Run-in Period: Placebo: Single-blind treatment with placebo for 14 to 17 days of the Screening period and before the first dose of double-blind study drug on Day 1.
- Double-Blind Treatment Period: Placebo 1; Double-Blind Treatment Period: IW-1701 (Olinciguat) 2 mg; Double-Blind Treatment Period: IW-1701 (Olinciguat) 6 mg: Participants receiving treatment under the original protocol, Amendment 1, Amendment 2, and Amendment 3
- Double-Blind Treatment Period: Placebo 2; Double-Blind Treatment Period: IW-1701 (Olinciguat) 18 mg: Participants receiving treatment under protocol Amendment 4 and later
- Double-Blind Treatment Period: IW-1701 (Olinciguat) 4 mg: Participants receiving treatment under the original protocol, Amendment 1, Amendment 2, and Amendment 3I
Arm/Group | Single-Blind Run-in Period: Placebo | Double-Blind Treatment Period: Placebo 1 | Double-Blind Treatment Period: Placebo 2 | Double-Blind Treatment Period: IW-1701 (Olinciguat) 2 mg | Double-Blind Treatment Period: IW-1701 (Olinciguat) 4 mg | Double-Blind Treatment Period: IW-1701 (Olinciguat) 6 mg | Double-Blind Treatment Period: IW-1701 (Olinciguat) 18 mg
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/9 | 0/8 | 0/8 | 0/8 | 0/11 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/88 | 2/9 | 1/8 | 2/8 | 3/8 | 4/11 | 6/24
Other Adverse Events (participants affected / at risk) | 18/88 | 6/9 | 6/8 | 5/8 | 5/8 | 6/11 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Blind Run-in Period: Placebo (N=88) | Double-Blind Treatment Period: Placebo 1 (N=9) | Double-Blind Treatment Period: Placebo 2 (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 2 mg (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 4 mg (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 6 mg (N=11) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 18 mg (N=24)
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 3 | 3 | 3
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Blind Run-in Period: Placebo (N=88) | Double-Blind Treatment Period: Placebo 1 (N=9) | Double-Blind Treatment Period: Placebo 2 (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 2 mg (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 4 mg (N=8) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 6 mg (N=11) | Double-Blind Treatment Period: IW-1701 (Olinciguat) 18 mg (N=24)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 2 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 2
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 5
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
GINGIVITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
SICKLE CELL ANAEMIA WITH CRISIS (Blood and lymphatic system disorders) | 3 | 1 | 1 | 3 | 1 | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 2 | 2
VOMITING (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 3
HEADACHE (Nervous system disorders) | 3 | 1 | 2 | 0 | 1 | 2 | 6
FATIGUE (General disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 2
SUPRAPUBIC PAIN (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
EARLY SATIETY (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VESSEL PUNCTURE SITE PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
INFUSION SITE EXTRAVASATION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
AMYLASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
MUMPS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL PAIN (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
PERIORBITAL SWELLING (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
GENITAL DISCOLOURATION (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
DEVICE MALFUNCTION (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03285178/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03285178/SAP_002.pdf